CLINICAL TRIAL: NCT02076074
Title: Evaluation of Single Fraction High-Gradient Partial Breast Irradiation as the Sole Method of Radiation Therapy for Low-Risk Stage 0 and I Breast Carcinoma
Brief Title: Single Fraction High-Gradient Partial Breast Irradiation in Treating Patients With Low-Risk Stage 0-I Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201401160
Record Dates: First submitted 2014-02-27; First posted 2014-03-03 (Estimated); Results first posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-06

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (HG-PBI) (Experimental): Patients undergo single fraction high gradient-partial breast irradiation within 8 weeks after partial mastectomy.
  Interventions: Radiation: accelerated partial breast irradiation

INTERVENTIONS:
Radiation: accelerated partial breast irradiation — Undergo HG-PBI
  Other Names: APBI

SUMMARY:
This phase I/II clinical trial studies the side effects of delivering radiation therapy in a single session instead of multiple treatments over several weeks and to see how well it works in treating patients with low-risk stage 0-I breast cancer. Partial-breast irradiation, a type of radiation therapy focused only to the part of the breast that has cancer in it, given at a lower dose than standard whole-breast radiation therapy. Single fraction high-gradient partial-breast irradiation may cause fewer side effects, help prevent breast cancer from coming back, and improve the appearance of the breast and quality of life of patients with breast cancer.

DETAILED DESCRIPTION:
This is a phase I/II study which will evaluate the complication rates, local control, cosmetic results, and quality of life of single fraction high gradient partial breast irradiation (HG-PBI) when used as the sole method of radiation therapy for patients with pathologic stage 0 (=< 2 cm) or I carcinoma of the breast treated with partial mastectomy with histologically assessed negative surgical margins.

ELIGIBILITY:
Inclusion Criteria:

* AJCC 7th Edition stage 0 or I (TisN0 ≤ 2 cm or T1N0) histologically confirmed carcinoma of the breast, treated with partial mastectomy. Axillary sampling is required only for cases of invasive cancers. Tumor size is determined by the pathologist. Clinical size may be used if the pathologic size is indeterminate. Patients with invasive cancer must have no positive axillary lymph nodes with at least 6 axillary lymph nodes sampled or a negative sentinel node.
* Negative histologic margins of partial mastectomy or re-excision specimen. Margins generally are positive if there is invasive or noninvasive tumor at the inked resection margin, close but negative if the tumor is within 2 mm of the inked margin and negative if the tumor is at least 2 mm away from the inked edge.
* Invasive ductal, lobular, medullary, papillary, colloid (mucinous), tubular histologies, or mixed histologies (lesions ≤ 2 cm) that are estrogen or progesterone receptor positive and do not exhibit HER2/neu gene amplification OR ductal carcinoma in situ (lesions ≤ 2 cm).
* Systemic therapy, if planned, must be adjuvant in nature and not be scheduled to begin for at least 4 weeks after completion of HG-PBI.
* Good candidate for treatment per protocol in the judgment of the PI and/or treating physician following simulation.
* Postmenopausal status.
* Age ≥ 50 years at diagnosis.
* Able to understand and willing to sign IRB-approved written informed consent document.
* English speaker.

Exclusion Criteria:

* Presence of distant metastases.
* In situ lobular carcinoma or nonepithelial breast malignancies such as sarcoma or lymphoma.
* Proven multicentric carcinoma (tumors in different quadrants of the breast, or tumors separated by at least 4 cm) with other clinically or radiographically suspicious areas in the ipsilateral breast unless confirmed to be negative for malignancy by biopsy.
* Premenopausal status.
* Histologically confirmed positive axillary nodes in the ipsilateral axilla. Palpable or radiographically suspicious contralateral axillary, supraclavicular, infraclavicular, or internal mammary nodes, unless there is histologic confirmation that these nodes are negative for tumor.
* Prior non-hormonal therapy for the present breast cancer, including radiation therapy or chemotherapy.
* Diagnosis of systemic lupus erythematosis, scleroderma, or dermatomyositis.
* Diagnosis of a coexisting medical condition which limits life expectancy to < 2 years.
* Diagnosis of psychiatric or addictive disorders that would preclude obtaining informed consent.
* History of other malignancy ≤ 5 years previous with the exception of basal cell or squamous cell carcinoma of the skin which were treated with local resection only or carcinoma in situ of the cervix.
* Paget's disease of the nipple.
* Skin involvement, regardless of tumor size.
* Unsatisfactory breast for HG-PBI as determined by the treating physician. For example, if there is little breast tissue remaining between the skin and pectoralis muscle after surgery, treatment with HG-PBI is technically problematic.
* Partial mastectomy so extensive that the cosmetic result is fair or poor prior to HG-PBI as determined by the treating physician.
* Surgical margins which cannot be microscopically assessed or are positive at pathological evaluation.
* Time between final definitive breast procedure to HG-PBI simulation is greater than 8 weeks.

Inclusion of Women and Minorities

-Women and members of all races and ethnic groups are eligible for this trial. Because breast cancer occurs rarely in men, men will not be recruited for participation.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-04-02 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2023-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Imran Zoberi, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (HG-PBI)
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (HG-PBI)
Number analyzed (Participants) | 50
Age, Continuous [Median (Full Range); unit: years] | 65 [52 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 48
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 44
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Are Free of Serious Treatment Related Toxicity
Description: Quantified by estimating the rate of acute and late treatment-related grade 3 or higher toxicity (per CTCAE, v.4.0) or any other grade 4 or 5 toxicity attributed to the therapy. Toxicities of concern include breast pain, delayed wound healing, persistent seroma fluid accumulation, breast fibrosis and fat necrosis in the treated breast. Rare toxicities include radiation pneumonitis and pericarditis. Acute toxicities are defined as toxicities that occurred from start of treatment until day 90. Late toxicities are defined as toxicities that occurred from Day 91 until completion of 5 year follow-up.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (HG-PBI)
Number analyzed (Participants) | 50
Participants
  Number of patients free of acute grade 3 or higher treatment related toxicity | 50
  Number of patients free of late grade 3 or higher treatment related toxicity | 49

2. Primary Outcome: Percentage of Patients Who Are Free of Breast Cancer in the Treated Breast
Description: Percentage of patients without ipsilateral breast tumor recurrences (IBTR).
Time Frame: At 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (HG-PBI)
Number analyzed (Participants) | 50
Participants | 48

3. Secondary Outcome: Percentage of Patients Who Are Free of Breast Cancer in the Regional Lymph Nodes
Description: Ipsilateral axilla, infraclavicular, supraclavicular, and internal mammary groups.
Time Frame: At 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (HG-PBI)
Number analyzed (Participants) | 50
Participants | 49

4. Secondary Outcome: Percentage of Patients Who Are Free From Distant Metastases
Time Frame: At 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (HG-PBI)
Number analyzed (Participants) | 50
Participants | 49

5. Secondary Outcome: Change in Quality of Life as Measured by the Mean Change From Baseline - EORTC QLC-C30
Description: The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale.
  All of the scales and single-item measures range in score from 0 to 100. For the global health and five functional scales (Cognitive Functioning, Emotional Functioning, Physical Functioning, Role Functioning, and Social Functioning) a high score correlates to a high level of functioning or a better outcome. For the three symptom scales and six single item scales (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Insomnia, Appetite loss, Constipation, Diarrhea, Financial Difficulties) a high score correlates to high levels of symptoms or problems and a worse outcome.
Time Frame: 2 weeks, 8 weeks, 6 months, 12 months, 18 months, 24 months, 36 months, year 4, and year 5
Population: If participants did not complete the questionnaire or did not complete a question then they are not included in the number analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Treatment (HG-PBI) - 2 Weeks; Treatment (HG-PBI) - 8 Weeks; Treatment (HG-PBI) - 6 Months; Treatment (HG-PBI) - 12 Months; Treatment (HG-PBI) - 18 Months; Treatment (HG-PBI) - 24 Months; Treatment (HG-PBI) - 36 Months; Treatment (HG-PBI) - Year 4; Treatment (HG-PBI) - Year 5: Patients undergo single fraction high gradient-partial breast irradiation within 8 weeks after partial mastectomy.
Arm/Group | Treatment (HG-PBI) - 2 Weeks | Treatment (HG-PBI) - 8 Weeks | Treatment (HG-PBI) - 6 Months | Treatment (HG-PBI) - 12 Months | Treatment (HG-PBI) - 18 Months | Treatment (HG-PBI) - 24 Months | Treatment (HG-PBI) - 36 Months | Treatment (HG-PBI) - Year 4 | Treatment (HG-PBI) - Year 5
Number analyzed (Participants) | 44 | 49 | 49 | 47 | 44 | 48 | 42 | 35 | 33
score on a scale
  Appetite Loss | -0.78 (15.41) | 0.68 (14.42) | 0.69 (12.84) | -1.42 (9.72) | 1.52 (14.3) | 2.08 (15.99) | -0.81 (11.76) | -1.9 (7.85) | 2.02 (8.08)
  Cognitive Functioning: number analyzed (Participants) | 44 | 49 | 49 | 47 | 43 | 48 | 42 | 34 | 32
  Cognitive Functioning | -2.27 (17.46) | -6.12 (18.22) | -6.46 (16.95) | -3.9 (16.74) | -5.43 (16.15) | -5.9 (13.96) | -1.59 (13.17) | -4.41 (12.52) | 0.52 (13.04)
  Constipation: number analyzed (Participants) | 44 | 49 | 49 | 47 | 43 | 48 | 42 | 34 | 32
  Constipation | 0 (20.33) | 0 (13.61) | 0.68 (14.42) | 1.42 (16.96) | 5.43 (26.16) | 1.39 (21.7) | -0.79 (11.61) | 0.98 (12.94) | 0 (20.74)
  Diarrhea: number analyzed (Participants) | 44 | 49 | 49 | 47 | 42 | 48 | 42 | 33 | 32
  Diarrhea | 0.76 (11.34) | 0 (15.21) | 0.68 (15.94) | -0.71 (8.48) | 0 (12.75) | 1.39 (13.68) | 2.38 (15.43) | 2.02 (16.54) | 1.04 (15.8)
  Dyspnea: number analyzed (Participants) | 43 | 49 | 49 | 47 | 44 | 48 | 41 | 35 | 33
  Dyspnea | -1.55 (19.18) | 1.36 (16.61) | 1.36 (13.54) | 5.67 (16.03) | 5.3 (18.94) | 8.33 (23.32) | 3.25 (10.01) | 3.81 (15.7) | 5.05 (18.86)
  Emotional Functioning: number analyzed (Participants) | 44 | 49 | 49 | 47 | 43 | 48 | 42 | 34 | 32
  Emotional Functioning | 1.07 (14.82) | 0.34 (15.31) | 1.93 (15.3) | 2.3 (15.22) | 4.52 (10.2) | 1.56 (16.09) | 0.79 (15.49) | 3.43 (11.07) | 4.25 (10.27)
  Fatigue | 5.68 (19.23) | 7.26 (13.38) | 3.51 (15.16) | 3.78 (15.59) | 1.64 (14.99) | 1.62 (16.04) | 0.4 (14.12) | 2.86 (16.47) | 5.05 (16.45)
  Financial Difficulties: number analyzed (Participants) | 41 | 46 | 46 | 44 | 40 | 45 | 39 | 32 | 29
  Financial Difficulties | 0.81 (26.34) | -0.72 (21.65) | -2.9 (19.66) | -6.06 (21.89) | -4.17 (18.78) | -1.48 (22.42) | -6.84 (19.01) | -5.21 (17.16) | -4.6 (14.7)
  Global Health Status: number analyzed (Participants) | 44 | 49 | 49 | 47 | 43 | 48 | 42 | 34 | 32
  Global Health Status | -0.57 (10.54) | -0.68 (8.81) | -2.89 (12.68) | -2.48 (12.76) | -4.26 (17.29) | -1.39 (15.21) | -3.57 (14.51) | -3.92 (17.44) | -1.3 (11.99)
  Insomnia: number analyzed (Participants) | 43 | 48 | 49 | 46 | 44 | 47 | 41 | 35 | 33
  Insomnia | -2.33 (23.45) | 3.47 (25.02) | 2.72 (33.22) | 2.17 (28.46) | -1.52 (28.71) | 5.67 (28.93) | 3.25 (29.63) | 5.71 (24.9) | 3.03 (24.1)
  Nausea and Vomiting: number analyzed (Participants) | 43 | 49 | 49 | 47 | 44 | 48 | 41 | 35 | 33
  Nausea and Vomiting | 2.71 (10.87) | 1.7 (7.01) | 1.36 (6.66) | 2.48 (10.41) | 3.79 (16.42) | 1.74 (7.87) | 0 (3.73) | 1.43 (7.42) | 0 (4.17)
  Pain: number analyzed (Participants) | 44 | 49 | 49 | 46 | 44 | 48 | 42 | 35 | 33
  Pain | -3.03 (18.42) | 0 (22.31) | -2.04 (20.59) | -3.26 (13.89) | -1.14 (18.47) | -1.39 (17.13) | -1.59 (23.52) | -3.81 (24.62) | -0.51 (23.01)
  Physical Functioning: number analyzed (Participants) | 43 | 49 | 49 | 47 | 44 | 48 | 42 | 35 | 33
  Physical Functioning | 0.67 (6.53) | -0.11 (11.19) | -1.58 (14.25) | -2.6 (11.59) | -0.66 (9.84) | -1.99 (12.58) | -1.63 (11.41) | -1.21 (10.62) | -2.79 (8.18)
  Role Functioning: number analyzed (Participants) | 43 | 49 | 49 | 47 | 44 | 48 | 42 | 35 | 33
  Role Functioning | 0 (23.85) | 0.68 (14.42) | 0.34 (12.02) | -0.35 (16.11) | 1.14 (14.56) | 1.74 (12.51) | -0.4 (16.66) | 0 (23.22) | -5.56 (20.27)
  Social Functioning: number analyzed (Participants) | 44 | 49 | 49 | 47 | 43 | 48 | 42 | 34 | 32
  Social Functioning | -1.14 (19.49) | 2.38 (11.28) | 2.38 (12.27) | 2.48 (14.74) | 4.26 (13.16) | 1.74 (15.47) | 1.98 (14.82) | 3.43 (14.67) | 4.69 (15.4)

6. Secondary Outcome: Change in Quality of Life as Measured by the Mean Change From Baseline - QLQ-BR23
Description: The QLQ-BR23 incorporates five multi-item scales to assess body image, sexual functioning, systemic therapy side effects, breast symptoms, and arm symptoms. In addition, single items assess sexual enjoyment, future perspective and being upset by hair loss.
  All of the scales and single-item measures range in score from 0 to 100. For the four symptom scales (Systemic Therapy Side Effects, Upset by Hair Loss, Arm Symptoms, Breast Symptoms) a high score correlates to high levels of symptoms or problems and a worse outcome. For the four functional scales (Body Image, Future Perspective, Sexual Functioning, Sexual Enjoyment) a high score correlates to a high/healthy level of functioning or a better outcome
Time Frame: 2 weeks, 8 weeks, 6 months, 12 months, 18 months, 24 months, 36 months, year 4, and year 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment (HG-PBI) - 2 Weeks | Treatment (HG-PBI) - 8 Weeks | Treatment (HG-PBI) - 6 Months | Treatment (HG-PBI) - 12 Months | Treatment (HG-PBI) - 18 Months | Treatment (HG-PBI) - 24 Months | Treatment (HG-PBI) - 36 Months | Treatment (HG-PBI) - Year 4 | Treatment (HG-PBI) - Year 5
Number analyzed (Participants) | 44 | 48 | 47 | 46 | 43 | 47 | 41 | 34 | 32
score on a scale
  Arm Symptoms | -2.02 (11.05) | -0.69 (12) | -0.47 (15.18) | -1.45 (11.14) | -3.23 (14.1) | -1.89 (12.33) | -3.52 (15.8) | -4.9 (18.59) | -2.08 (11.79)
  Body Image: number analyzed (Participants) | 42 | 47 | 46 | 45 | 43 | 46 | 40 | 34 | 31
  Body Image | 2.31 (10.32) | 1.6 (8.97) | 0 (7.66) | -0.37 (10.65) | 1.23 (10.49) | 0.66 (9.45) | -0.9 (13.17) | -0.98 (14.76) | -1.61 (12.98)
  Breast Symptoms | -1.83 (11.54) | -3.3 (15.54) | -6.86 (14.74) | -8.76 (10.44) | -10.08 (11.72) | -9.63 (13.57) | -11.04 (11.94) | -8.25 (11.16) | -8.94 (10.65)
  Future Perspective: number analyzed (Participants) | 42 | 47 | 46 | 45 | 43 | 46 | 40 | 34 | 32
  Future Perspective | -3.97 (18.34) | -4.96 (25.04) | -2.17 (23.73) | -7.41 (24.5) | -6.2 (31.92) | -4.35 (23.94) | -7.5 (26.67) | -11.76 (29.45) | -10.75 (29.04)
  Sexual Enjoyment: number analyzed (Participants) | 14 | 14 | 12 | 15 | 12 | 13 | 11 | 7 | 6
  Sexual Enjoyment | 2.38 (15.82) | 4.76 (25.68) | -2.78 (26.43) | 0 (21.82) | 5.56 (19.25) | 2.56 (21.35) | 9.09 (30.15) | -4.76 (12.6) | -5.56 (13.61)
  Sexual Functioning: number analyzed (Participants) | 41 | 46 | 43 | 42 | 40 | 43 | 37 | 29 | 28
  Sexual Functioning | -4.88 (17.18) | -4.35 (17.72) | -3.88 (14.01) | -5.16 (15.39) | -7.5 (14.1) | -0.39 (19.41) | -5.41 (19.66) | -4.02 (23.42) | -1.19 (21.24)
  Systemic Therapy Side Effects: number analyzed (Participants) | 43 | 48 | 47 | 46 | 43 | 47 | 41 | 34 | 32
  Systemic Therapy Side Effects | 3.7 (10.3) | 7.75 (10.76) | 8.1 (11.46) | 5.13 (12.22) | 3.75 (8.71) | 4.67 (10.26) | 2.72 (7.71) | 2.5 (7.02) | 3.14 (10.38)
  Upset by Hair Loss: number analyzed (Participants) | 1 | 4 | 5 | 5 | 3 | 4 | 3 | 2 | 2
  Upset by Hair Loss | 33.33 (NA) — There was only one participant evaluable so SD is not available. | 16.67 (33.33) | -26.67 (43.46) | -20 (29.81) | 0 (0) | 0 (27.22) | -44.44 (38.49) | 0 (0) | -50 (23.57)

7. Secondary Outcome: Change in Quality of Life as Measured by the Mean Change From Baseline - Visual Analog Scale for Pain
Description: The pain VAS is a unidimensional measure of pain intensity, used to record patients' pain progression, or compare pain severity between patients with similar conditions. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor (0) and "severe pain" at (10) with the patient's mark providing a range of scores from 0-100 millimeters. A higher score indicates greater pain intensity.
Time Frame: 2 weeks, 8 weeks, 6 months, 12 months, 18 months, 24 months, 36 months, year 4, and year 5
Population: If participants did not complete the questionnaire then they are not included in the number analyzed.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Treatment (HG-PBI) - 2 Weeks | Treatment (HG-PBI) - 8 Weeks | Treatment (HG-PBI) - 6 Months | Treatment (HG-PBI) - 12 Months | Treatment (HG-PBI) - 18 Months | Treatment (HG-PBI) - 24 Months | Treatment (HG-PBI) - 36 Months | Treatment (HG-PBI) - Year 4 | Treatment (HG-PBI) - Year 5
Number analyzed (Participants) | 41 | 49 | 47 | 44 | 42 | 49 | 39 | 35 | 31
mm | -0.34 (0.94) | -0.14 (1.29) | -0.43 (1.44) | -0.59 (1.23) | -0.67 (1.49) | -0.63 (1.51) | -0.62 (1.14) | -0.6 (1.29) | -0.74 (1.03)

8. Secondary Outcome: Cosmesis as Measured by the Mean Change From Baseline - Breast Retraction Assessment (BRA)
Description: This instrument includes a formula expressing the extent of displacement of the treated breast relative to the contralateral breast and other anatomical features.
Time Frame: 8 weeks, 6 months, 12 months, 24 months, 36 months, year 4, and year 5
Population: If participants missed the BRA then they are not included in the number analyzed.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Treatment (HG-PBI) - 8 Weeks | Treatment (HG-PBI) - 6 Months | Treatment (HG-PBI) - 12 Months | Treatment (HG-PBI) - 24 Months | Treatment (HG-PBI) - 36 Months | Treatment (HG-PBI) - Year 4 | Treatment (HG-PBI) - Year 5
Number analyzed (Participants) | 49 | 47 | 46 | 42 | 37 | 33 | 27
cm | -0.14 (1.08) | 0.22 (3.41) | -0.15 (2.89) | -0.5 (1.08) | 0.21 (3.09) | 0.34 (4.08) | 0.91 (4.85)

9. Secondary Outcome: Cosmesis as Measured by the Mean Change From Baseline - Percentage Breast Retraction Assessment (pBRA)
Description: This instrument includes a formula expressing the extent of displacement of the treated breast relative to the contralateral breast and other anatomical features. This is calculated from dividing the BRA score by the reference length from sternal notch to contralateral nipple and then multiplying that value by 100 to get a percentage.
Time Frame: 8 weeks, 6 months, 12 months, 24 months, 36 months, year 4, and year 5
Population: If participants did not have the percentage Breast Retraction Assessment then they are not included in the analysis.
Measure: Mean (Standard Deviation); unit: percentage breast retraction
Arm/Group | Treatment (HG-PBI) - 8 Weeks | Treatment (HG-PBI) - 6 Months | Treatment (HG-PBI) - 12 Months | Treatment (HG-PBI) - 24 Months | Treatment (HG-PBI) - 36 Months | Treatment (HG-PBI) - Year 4 | Treatment (HG-PBI) - Year 5
Number analyzed (Participants) | 48 | 47 | 44 | 43 | 35 | 31 | 28
percentage breast retraction | -1.05 (5.14) | -0.67 (10.37) | -1.81 (9.71) | -2.93 (5.24) | -1.76 (9.2) | -1.56 (11.29) | -0.03 (14.29)

10. Secondary Outcome: Cosmesis as Measured by the Mean Change From Baseline - Aronson Modified Harris Scale.
Description: Using this scale, cosmesis is qualitatively evaluated by the treating radiation oncologist by comparing the treated breast with the contralateral breast using the Aronson Modified Scale. The global cosmetic result, appearance of the surgical scar, breast size, breast shape, skin color, location of the areola and nipple, and shape of the areola and nipple were scored on a 4-point scale. In this case 1 is 'excellent' with 4 being 'poor.'
Time Frame: 8 weeks, 6 months, 12 months, 24 months, 36 months, year 4, and year 5
Population: If physicians did not complete the evaluation with the participant then they are not included in the number analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment (HG-PBI) - 8 Weeks | Treatment (HG-PBI) - 6 Months | Treatment (HG-PBI) - 12 Months | Treatment (HG-PBI) - 18 Months | Treatment (HG-PBI) - 24 Months | Treatment (HG-PBI) - 36 Months | Treatment (HG-PBI) - Year 4 | Treatment (HG-PBI) - Year 5
Number analyzed (Participants) | 47 | 47 | 44 | 38 | 42 | 37 | 33 | 29
score on a scale | -0.04 (0.36) | -0.09 (0.28) | 0.02 (0.4) | 0.03 (0.37) | 0 (0.31) | 0.05 (0.4) | 0.09 (0.58) | 0.21 (0.49)

11. Secondary Outcome: Number of Patients With Complications Using CTCAE v. 4.0
Description: Acute complications are defined as complications that occurred from start of treatment until day 90. Late complications are defined as complications that occurred from Day 91 until completion of 5 year follow-up.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Groups:
- Treatment (HG-PBI) - Acute; Treatment (HG-PBI) - Late: Patients undergo single fraction high gradient-partial breast irradiation within 8 weeks after partial mastectomy.
Arm/Group | Treatment (HG-PBI) - Acute | Treatment (HG-PBI) - Late
Number analyzed (Participants) | 50 | 50
Participants
  Alkaline phosphatase increased | 0 | 1
  Alopecia | 3 | 3
  Anemia | 0 | 2
  Arthralgia | 6 | 30
  Ataxia | 0 | 1
  Atrial Fibrillation | 0 | 1
  Back Pain | 1 | 4
  Breast Atrophy | 0 | 1
  Breast Pain | 3 | 7
  Bronchial Infection | 0 | 1
  Congestive heart failure | 0 | 1
  Chest pain - Cardiac | 0 | 1
  Chest Wall Pain | 1 | 0
  Chills | 0 | 1
  Chronic kidney disease | 0 | 1
  Constipation | 0 | 1
  Cough | 0 | 1
  Depression | 0 | 1
  Diarrhea | 0 | 1
  Dizziness | 0 | 1
  Dry Mouth | 0 | 2
  Dry Skin | 0 | 1
  Dyspnea | 0 | 4
  Edema Limbs | 0 | 3
  Ejection fraction decreased | 0 | 1
  Epistaxis | 0 | 1
  Fall | 0 | 2
  Fatigue | 2 | 4
  Fibrosis deep connective tissue | 1 | 24
  Flank Pain | 0 | 1
  Gastroesophageal reflux disease | 1 | 1
  Poor dentition | 0 | 1
  Headache | 1 | 0
  Heart Failure | 0 | 1
  Hematoma | 0 | 1
  Hot Flashes | 13 | 34
  Hyperhidrosis | 10 | 22
  Hyperkalemia | 0 | 1
  Hypertension | 0 | 1
  Candida infection | 0 | 1
  COVID-19 infection | 0 | 1
  Insomnia | 0 | 3
  Irritability | 0 | 1
  Joint infection | 0 | 1
  Memory Impairment | 0 | 3
  Shoulder pain | 1 | 0
  Myocardial Infarction | 0 | 1
  Nausea | 1 | 0
  Neck Pain | 0 | 2
  Neutrophil Count Decreased | 0 | 1
  Nipple deformity | 0 | 1
  Pain in extremity | 0 | 1
  Pain | 1 | 0
  Pericardial Effusion | 0 | 1
  Platelet Count decrease | 0 | 1
  Seroma | 3 | 1
  Skin Atrophy | 0 | 5
  Skin Hyperpigmentation | 15 | 16
  Skin Induration | 1 | 4
  Skin Infection | 0 | 1
  Superficial soft tissue fibrosis | 3 | 7
  Telangiectasia | 0 | 1
  Thrombotic event | 0 | 1
  Tremor | 0 | 1
  Upper respiratory Infection | 1 | 1
  Urticaria | 1 | 0
  Vaginal Pain | 0 | 1
  Vertigo | 0 | 1
  Vomiting | 1 | 0
  White blood cell decrease | 0 | 1
  Shingles | 0 | 1
  Scar retraction | 0 | 1
  Trigger finger | 0 | 1

12. Secondary Outcome: Number of Participants With Grade 3-4 Toxicities Using CTCAE v4.0
Description: Acute toxicities are defined as toxicities that occurred from start of treatment until day 90. Late toxicities are defined as toxicities that occurred from Day 91 until completion of 5 year follow-up.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (HG-PBI)
Number analyzed (Participants) | 50
Participants
  Late - fibrosis deep connective tissue | 1
  Late - neutrophil count decreased | 1
  Late - white blood cell decreased | 1

13. Secondary Outcome: Percentage of Patients Undergoing Mastectomy on the Treated Side
Time Frame: At 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (HG-PBI)
Number analyzed (Participants) | 50
Participants | 1

ADVERSE EVENTS:
Time Frame: Adverse events and all-cause mortality was collected from start of treatment through completion of follow-up (up to 5 years).
Description: Acute adverse events are defined as adverse events that occurred from start of treatment until day 90. Late adverse events are defined as adverse events that occurred from Day 91 until completion of 5 year follow-up.
Arm/Group | Treatment (HG-PBI) - Acute | Treatment (HG-PBI) - Late
All-Cause Mortality (participants affected / at risk) | 0/50 | 4/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 32/50 | 48/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (HG-PBI) - Acute (N=50) | Treatment (HG-PBI) - Late (N=50)
Anemia (Blood and lymphatic system disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 1
Chest pain - cardiac (Cardiac disorders) | 0 | 1
Congestive heart failure (Cardiac disorders) | 0 | 1
Heart failure (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Poor dentition (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Chills (General disorders) | 0 | 1
Edema limbs (General disorders) | 0 | 3
Fatigue (General disorders) | 2 | 4
Pain (General disorders) | 1 | 0
Pain in extremity (General disorders) | 0 | 1
Bronchial infection (Infections and infestations) | 0 | 1
COVID-19 infection (Infections and infestations) | 0 | 1
Candida infection (Infections and infestations) | 0 | 1
Joint infection (Infections and infestations) | 0 | 1
Shingles (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Upper respiratory infection (Infections and infestations) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 2
Scar retraction (Injury, poisoning and procedural complications) | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 3 | 1
Alkaline phosphatase increased (Investigations) | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
White blood cell decreased (Investigations) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 30
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 4
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Fibrosis deep connective tissue (Musculoskeletal and connective tissue disorders) | 1 | 24
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Superficial soft tissue fibrosis (Musculoskeletal and connective tissue disorders) | 3 | 7
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 1
Ataxia (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 3
Tremor (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 3
Irritability (Psychiatric disorders) | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 1
Breast atrophy (Reproductive system and breast disorders) | 0 | 1
Breast pain (Reproductive system and breast disorders) | 3 | 7
Nipple deformity (Reproductive system and breast disorders) | 0 | 1
Vaginal pain (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 10 | 22
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 | 5
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 15 | 16
Skin induration (Skin and subcutaneous tissue disorders) | 1 | 4
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Hematoma (Vascular disorders) | 0 | 1
Hot flashes (Vascular disorders) | 13 | 34
Hypertension (Vascular disorders) | 0 | 1
Thrombotic event (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-26): https://cdn.clinicaltrials.gov/large-docs/74/NCT02076074/Prot_SAP_000.pdf